CLINICAL TRIAL: NCT03840148
Title: A Phase 3, Randomized, Double-blind, Active Controlled Noninferiority Study Evaluating the Efficacy, Safety, and Tolerability of Cefepime/VNRX-5133 in Adults With Complicated Urinary Tract Infections (cUTI), Including Acute Pyelonephritis
Brief Title: Safety and Efficacy Study of Cefepime/VNRX-5133 in Patients With Complicated Urinary Tract Infections
Acronym: CERTAIN-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Venatorx Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VNRX-5133-201; 2018-001451-13 (EudraCT Number)
Record Dates: First submitted 2019-02-06; First posted 2019-02-15 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Urinary Tract Infections; Acute Pyelonephritis
Keywords: Bacterial Infections; Cefepime; Meropenem; Complicated Urinary Tract Infections; Anti-Infective Agents; β-Lactamase Inhibitors; VNRX-5133 (taniborbactam)
MeSH Terms: conditions — Urinary Tract Infections; Bacterial Infections | interventions — taniborbactam; Meropenem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cefepime/VNRX-5133 (taniborbactam) (Experimental): Cefepime/VNRX-5133 administered q8h intravenously (IV) over a 2-hour period.
  Interventions: Drug: Cefepime/VNRX-5133 (taniborbactam)
- Meropenem (Active Comparator): Meropenem will be administered q8h IV over 30 minutes.
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Cefepime/VNRX-5133 (taniborbactam) — Cefepime/VNRX-5133 administered q8h intravenously (IV) over a 2-hour period for 7 days (up to 14 days for patients with bacteremia). Patients will also receive meropenem placebo administered via IV over 30 minutes.
  Arms: Cefepime/VNRX-5133 (taniborbactam)
Drug: Meropenem — Meropenem will be administered q8h IV over 30 minutes for 7 days (up to 14 days for patients with bacteremia). Patients will also receive cefepime/VNRX-5133 placebo administered via IV over a 2-hour period.
  Arms: Meropenem

SUMMARY:
This study will assess the safety and efficacy of cefepime/VNRX-5133 compared with meropenem in both eradication of bacteria and in symptomatic response in patients with cUTIs.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female
* Documented diagnosis of pyuria
* Documented diagnosis of cUTI or Acute Pyelonephritis (AP)

Exclusion Criteria:

* Receipt of effective antibacterial drug therapy for cUTI for more than 24 hours during the previous 72 hours prior to randomization
* A urine culture result is resistant to meropenem or a gram negative pathogen is not identified or more than 2 microorganisms are isolated or a confirmed fungal UTI is identified
* Required use of nonstudy systemic bacterial therapy
* Suspected or confirmed prostatitis or urinary tract symptoms attributable to sexually transmitted disease
* Patients with perinephric or renal abscess
* Patients with renal transplantation or receiving hemodialysis or peritoneal dialysis
* Abnormal labs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (78):
- United States (4):
  - Site 184003, Buena Park, California
  - Site 184002, Chula Vista, California
  - Site 184001, La Mesa, California
  - 184012, Northridge, California
- Site 103203, Córdoba, Argentina
- Brazil (2):
  - Site 107601, Belo Horizonte
  - Site 107608, São Paulo
- Bulgaria (9):
  - Site 110009, Gabrovo
  - Site 110002, Pleven
  - Site 110007, Plovdiv
  - Site 110003, Rousse
  - Site 110010, Sofia
  - Site 110004, Sofia
  - Site 110005, Sofia
  - Site 110008, Sofia
  - Site 110001, Veliko Tarnovo
- China (23):
  - Site 156022, Baotou
  - Site 156002, Beijing
  - Site 156006, Beijing
  - Site 156015, Chendu
  - Site 156011, Chongqing
  - Site 156012, Chongqing
  - Site 156004, Dalian
  - Site 156030, Fujian
  - Site 156014, Guangdong
  - Site 156027, Guangdong
  - Site 156025, Guangzhou
  - Site 156018, Guiyang
  - Site 156003, Nanchang
  - Site 156005, Nanjing
  - Site 156008, Nanjing
  - Site 156007, Nanjing
  - Site 156013, Ningbo
  - Site 156028, Shandong
  - Site 156017, Shanghai
  - Site 156016, Shijiazhuang
  - Site 156020, Tianjin
  - Site 156029, Ürümqi
  - Site 156010, Xiamen
- Croatia (3):
  - Site 119103, Split
  - Site 119101, Zagreb
  - Site 119106, Zagreb
- Hungary (3):
  - Site 134801, Budapest
  - Site 134803, Nyíregyháza
  - Site 134804, Szeged
- Latvia (3):
  - Site 142803, Daugavpils
  - Site 142804, Riga
  - Site 142801, Riga
- Mexico (2):
  - Site 148402, Colima
  - Site 148401, Guadalajara
- Peru (4):
  - Site 160403, Cuzco
  - Site 160410, Lima
  - Site 160406, Lima
  - Site 160404, Trujillo
- Romania (4):
  - Site 164206, Bucharest
  - Site 164205, Bucharest
  - Site 164204, Bucharest
  - Site 164201, Craiova
- Russia (6):
  - Site 164307, Moscow
  - Site 164301, Penza
  - Site 164308, Pyatigorsk
  - Site 164311, Rostov-on-Don
  - Site 164303, Saint Petersburg
  - Site 164302, Saratov
- Serbia (2):
  - Site 189001, Belgrade
  - Site 189002, Belgrade
- Turkey (Türkiye) (5):
  - Site 179207, Adapazarı
  - Site 179203, Bornova
  - Site 179202, Bostancı
  - Site 179205, Çankaya
  - Site 179204, Diyarbakır
- Ukraine (7):
  - Site 180404, Dnipro
  - Site 180408, Ivano-Frankivsk
  - Site 180402, Kharkiv
  - Site 180406, Kyiv
  - Site 180401, Lutsk
  - Site 180403, Vinnytsia
  - Site 180407, Zaporizhzhya

REFERENCES:
- [Derived] Moeck G, Gasink LB, Mendes RE, Woosley LN, Dorr M, Chen H, Wagenlehner FM, Henkel T, McGovern PC. Patient outcomes by baseline pathogen resistance phenotype and genotype in CERTAIN-1, a Phase 3 study of cefepime-taniborbactam versus meropenem in adults with complicated urinary tract infection. Antimicrob Agents Chemother. 2024 Jul 9;68(7):e0023624. doi: 10.1128/aac.00236-24. Epub 2024 May 23. PMID 38780262
- [Derived] Wagenlehner FM, Gasink LB, McGovern PC, Moeck G, McLeroth P, Dorr M, Dane A, Henkel T; CERTAIN-1 Study Team. Cefepime-Taniborbactam in Complicated Urinary Tract Infection. N Engl J Med. 2024 Feb 15;390(7):611-622. doi: 10.1056/NEJMoa2304748. PMID 38354140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six-hundred sixty-one (661) male and female patients with complicated urinary tract infection (cUTI) including acute pyelonephritis (AP), were randomized into 2 groups (cefepime - VNRX-5133, and meropenem) at 68 hospital sites in North and South America, Eastern Europe, and China, from August 2019 until the last patient's final visit in December 2021. Of these 661 patients in the intent-to-treat (ITT) population, 436 were in the MicroITT population (293 cefepime - VNRX-5133, 143 meropenem).
Pre-assignment Details: Of the 697 patients screened, 36 patients did not qualify for randomization, and 661 patients were randomized into the trial.
Period: Study Drug Disposition
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Started | 441 | 220
Completed (Randomized patients that completed study drug treatment.) | 414 | 212
Not Completed | 27 | 8
Not completed — Adverse Event | 13 | 2
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Lack of Efficacy | 3 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Randomized but not treated, IWRS issue, lack of IMP supplies. | 1 | 4
Period: Study Completion Disposition
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Started (The patients in this period are inclusive of those patients that either completed or did not complete the Study Drug Disposition period.) | 441 | 220
Completed (Randomized patients that completed the Late Follow-up Visit.) | 426 | 214
Not Completed | 15 | 6
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Covid-19 related | 2 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 1 | 0
Not completed — IWRS issue, patient refused, SAE, randomized in error, patient did not take IMP or attend visits. | 3 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem | Total
Number analyzed (Participants) | 441 | 220 | 661
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (17.43) | 55.8 (18.15) | 56.1 (17.66)
Age, Customized [Count of Participants; unit: Participants]
  Age Categories (years): <65 | 275 | 137 | 412
  Age Categories (years): 65 - 75 | 111 | 56 | 167
  Age Categories (years): >75 | 55 | 27 | 82
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 115 | 363
  Male | 193 | 105 | 298
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 20 | 67
  Not Hispanic or Latino | 393 | 199 | 592
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — The 12 participants in the cefepime/VNRX-5133 treatment arm and 8 in the meropenem treatment arm classified as "Unknown or Not Reported", were identified in the trial as "Other".
  Participants
    American Indian or Alaska Native | 4 | 1 | 5
    Asian | 36 | 17 | 53
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 3 | 6
    White | 386 | 191 | 577
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Composite Success at Test of Cure (TOC) in the Microbiological Intent-to-treat (microITT) Population
Description: Microbiologic success is eradication defined as demonstration that any gram-negative bacterial pathogen found at study entry (≥10^5 CFU/mL) is eradicated to <10^3 CFU/mL. Clinical success is defined as symptomatic resolution or return to pre-morbid baseline of all UTI-core symptoms and patient is alive, and patient has not received additional antibacterial therapy for cUTI.
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: The microITT analysis population consists of all patients in the ITT analysis population who had a positive study entry urine culture defined as ≥10^5 CFU/mL of a gram-negative pathogen(s) against which both cefepime/VNRX-5133 and meropenem have antibacterial activity AND those patients who had no more than 2 microorganisms identified in the study entry culture regardless of colony count.
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 293 | 143
Participants | 207 | 83
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Non-Inferiority — If the lower limit of the 95% CI for the difference in response is greater than or equal to the non-inferiority margin of -15%, non-inferiority will be concluded. Further, if non-inferiority is concluded, superiority will be concluded if the lower limit of the 95% CI for the difference in response is greater than or equal to zero; p = 0.0088, Cochran-Mantel-Haenszel — P-value for superiority since the lower confidence interval is greater than 0 for the primary endpoint analysis; Miettinen and Nurminen = 12.6, 95% CI 2-sided [3.1 to 22.2]

2. Secondary Outcome: Microbiologic Success at Test of Cure (TOC) in the microITT Population
Description: Microbiologic success is eradication defined as demonstration that any gram-negative bacterial pathogen found at study entry (≥10^5 CFU/mL) is eradicated to <10^3 CFU/mL.
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 293 | 143
Participants | 229 | 95
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 11.7, 95% CI 2-sided [2.9 to 21.0]

3. Secondary Outcome: Clinical Success at Test of Cure (TOC) in the microITT Population
Description: Symptomatic resolution or return to pre-morbid baseline of all UTI-core symptoms and patient is alive, and patient has not received additional antibacterial therapy for cUTI.
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 293 | 143
Participants | 251 | 116
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 4.5, 95% CI 2-sided [-2.6 to 12.6]

4. Secondary Outcome: Composite Success at Test of Cure (TOC) in the Extended Microbiological Intent-to-treat (emicroITT) Population
Description: Microbiologic success is eradication defined as demonstration that any gram-negative bacterial pathogen found at study entry (≥10^5 CFU/mL) is eradicated to <10^3 CFU/mL. Symptomatic clinical success is defined as symptomatic resolution or return to pre-morbid baseline of all UTI-core symptoms and patient is alive, and patient has not received additional antibacterial therapy for cUTI.
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: The extended microITT analysis population consists of all patients in the ITT analysis population who had a positive study entry urine culture defined as ≥10^5 CFU/mL of a gram-negative pathogen(s) against which at least 1 study drug (cefepime/VNRX-5133 and/or meropenem) have antibacterial activity AND those patients who had no more than 2 microorganisms identified in the study entry culture regardless of colony count.
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 305 | 147
Participants | 216 | 86
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 12.3, 95% CI 2-sided [3.0 to 21.8]

5. Secondary Outcome: Composite Success at End of Treatment (EOT) in the microITT Population
Description: as for outcome 1
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 293 | 143
Participants | 261 | 123
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 3.1, 95% CI 2-sided [-3.2 to 10.4]

6. Secondary Outcome: Microbiological Success at End of Treatment (EOT) in the microITT Population
Description: as for outcome 2
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 293 | 143
Participants | 284 | 139
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = -0.3, 95% CI 2-sided [-3.5 to 4.1]

7. Secondary Outcome: Clinical Success at End of Treatment (EOT) in the microITT Population
Description: Clinical success is defined as symptomatic resolution or return to pre-morbid baseline of all UTI-core symptoms and patient is alive, and patient has not received additional antibacterial therapy for cUTI.
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 293 | 143
Participants | 265 | 127
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 1.6, 95% CI 2-sided [-4.1 to 8.5]

8. Secondary Outcome: Composite Success at Late Follow Up (LFU) in the microITT Population
Description: as for outcome 1
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 293 | 143
Participants | 187 | 74
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 12.1, 95% CI 2-sided [2.2 to 21.9]

9. Secondary Outcome: Microbiological Success at Late Follow Up (LFU) in the microITT Population
Description: as for outcome 2
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 293 | 143
Participants | 207 | 90
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 7.7, 95% CI 2-sided [-1.6 to 17.3]

10. Secondary Outcome: Clinical Success at Late Follow Up (LFU) in the microITT Population
Description: as for outcome 7
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 293 | 143
Participants | 238 | 102
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 9.9, 95% CI 2-sided [1.5 to 18.8]

11. Secondary Outcome: Investigator Opinion of Clinical Success at Test of Cure (TOC) in the microITT Population
Description: The proportion of patients with clinical success based on investigator opinion at TOC.
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 293 | 143
Participants | 271 | 128
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 3.0, 95% CI 2-sided [-2.4 to 9.6]

12. Secondary Outcome: Composite Success in Patients With Cefepime-Resistant Pathogens at End of Treatment (EOT) in the microITT Population
Description: as for outcome 1
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 67 | 30
Participants
  Cefepime-resistant Enterobacterales: number analyzed (Participants) | 66 | 30
  Cefepime-resistant Enterobacterales | 57 | 26
  Cefepime-resistant Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Cefepime-resistant Pseudomonas aeruginosa | 1 |

13. Secondary Outcome: Microbiologic Success in Patients With Cefepime-Resistant Pathogens at End of Treatment (EOT) in the microITT Population
Description: as for outcome 2
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 67 | 30
Participants
  Cefepime-resistant Enterobacterales: number analyzed (Participants) | 66 | 30
  Cefepime-resistant Enterobacterales | 65 | 28
  Cefepime-resistant Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Cefepime-resistant Pseudomonas aeruginosa | 1 |

14. Secondary Outcome: Clinical Success in Patients With Cefepime-Resistant Pathogens at End of Treatment (EOT) in the microITT Population
Description: as for outcome 7
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 67 | 30
Participants
  Enterobacterales: number analyzed (Participants) | 66 | 30
  Enterobacterales | 57 | 28
  Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Pseudomonas aeruginosa | 1 |

15. Secondary Outcome: Composite Success in Patients With Cefepime-Resistant Pathogens at Test of Cure (TOC) in the microITT Population
Description: as for outcome 1
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 67 | 30
Participants
  Cefepime-resistant Enterobacterales: number analyzed (Participants) | 66 | 30
  Cefepime-resistant Enterobacterales | 47 | 16
  Cefepime-resistant Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Cefepime-resistant Pseudomonas aeruginosa | 0 |

16. Secondary Outcome: Microbiologic Success in Patients With Cefepime-Resistant Pathogens at Test of Cure (TOC) in the microITT Population
Description: as for outcome 2
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 67 | 30
Participants
  Cefepime-resistant Enterobacterales: number analyzed (Participants) | 66 | 30
  Cefepime-resistant Enterobacterales | 50 | 18
  Cefepime-resistant Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Cefepime-resistant Pseudomonas aeruginosa | 0 |

17. Secondary Outcome: Clinical Success in Patients With Cefepime-Resistant Pathogens at Test of Cure (TOC) in the microITT Population
Description: as for outcome 7
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 67 | 30
Participants
  Enterbacterales: number analyzed (Participants) | 66 | 30
  Enterbacterales | 54 | 25
  Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Pseudomonas aeruginosa | 0 |

18. Secondary Outcome: Composite Success in Patients With Cefepime-Resistant Pathogens at Late Follow Up (LFU) in the microITT Population
Description: as for outcome 1
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 67 | 30
Participants
  Cefepime-resistant Enterobacterales: number analyzed (Participants) | 66 | 30
  Cefepime-resistant Enterobacterales | 45 | 13
  Cefepime-resistant Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Cefepime-resistant Pseudomonas aeruginosa | 0 |

19. Secondary Outcome: Microbiologic Success in Patients With Cefepime-Resistant Pathogens at Late Follow Up (LFU) in the microITT Population
Description: as for outcome 2
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 67 | 30
Participants
  Cefepime-resistant Enterobacterales: number analyzed (Participants) | 66 | 30
  Cefepime-resistant Enterobacterales | 48 | 16
  Cefepime-resistant Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Cefepime-resistant Pseudomonas aeruginosa | 0 |

20. Secondary Outcome: Clinical Success in Patients With Cefepime-Resistant Pathogens at Late Follow Up (LFU) in the microITT Population
Description: as for outcome 7
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 67 | 30
Participants
  Enterobacterales: number analyzed (Participants) | 66 | 30
  Enterobacterales | 49 | 20
  Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Pseudomonas aeruginosa | 0 |

21. Secondary Outcome: Composite Success at End of Treatment (EOT) in the Microbiologically-Evaluable (ME) Population
Description: as for outcome 1
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: All patients who meet the criteria for the microITT population AND had a diagnosis of cUTI; received treatment for ≥48 hours; were evaluated at EOT with a response that was not indeterminate; did not violate prior antibacterials exclusion or received concomitant antibiotic therapy with activity against baseline pathogens except for patients failing study drug; or had other confounding factors that interfered with the assessment of outcome including unblinding.
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 282 | 137
Participants | 259 | 121
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 3.5, 95% CI 2-sided [-2.3 to 10.5]

22. Secondary Outcome: Microbiologic Success at End of Treatment (EOT) in the ME Population
Description: as for outcome 2
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 282 | 137
Participants | 279 | 137
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = -1.1, 95% CI 2-sided [-3.1 to 1.7]

23. Secondary Outcome: Composite Success at Test of Cure (TOC) in the ME Population
Description: as for outcome 4
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: All patients who meet the criteria for the microITT population AND had a diagnosis of cUTI; received treatment for ≥48 hours; were evaluated at TOC with a response that was not indeterminate; did not violate prior antibacterials exclusion or received concomitant antibiotic therapy with activity against baseline pathogens except for patients failing study drug; or had other confounding factors that interfered with the assessment of outcome including unblinding.
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 261 | 127
Participants | 195 | 76
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 14.9, 95% CI 2-sided [5.0 to 24.9]

24. Secondary Outcome: Microbiologic Success at Test of Cure (TOC) in the ME Population
Description: as for outcome 2
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 261 | 127
Participants | 214 | 88
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 12.7, 95% CI 2-sided [3.7 to 22.3]

25. Secondary Outcome: Composite Success at Late Follow Up (LFU) in the ME Population
Description: as for outcome 4
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: All patients who meet the criteria for the microITT population AND had a diagnosis of cUTI; received treatment for ≥48 hours; were evaluated at LFU with a response that was not indeterminate; did not violate prior antibacterials exclusion or received concomitant antibiotic therapy with activity against baseline pathogens except for patients failing study drug; or had other confounding factors that interfered with the assessment of outcome including unblinding.
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 262 | 128
Participants | 178 | 69
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 14.0, 95% CI 2-sided [3.8 to 24.3]

26. Secondary Outcome: Microbiologic Success at Late Follow Up (LFU) in the ME Population
Description: as for outcome 2
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 262 | 128
Participants | 192 | 84
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 7.7, 95% CI 2-sided [-1.9 to 17.7]

27. Secondary Outcome: Composite Success in Patients With Cefepime-Resistant Pathogens at the End of Treatment (EOT) in the ME Population
Description: as for outcome 4
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 64 | 28
Participants
  Cefepime-resistant Enterobacterales: number analyzed (Participants) | 63 | 28
  Cefepime-resistant Enterobacterales | 56 | 26
  Cefepime-resistant Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Cefepime-resistant Pseudomonas aeruginosa | 1 |

28. Secondary Outcome: Microbiologic Success in Patients With Cefepime-Resistant Pathogens at the End of Treatment (EOT) in the ME Population
Description: as for outcome 2
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 64 | 28
Participants
  Cefepime-resistant Enterobacterales: number analyzed (Participants) | 63 | 28
  Cefepime-resistant Enterobacterales | 62 | 28
  Cefepime-resistant Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Cefepime-resistant Pseudomonas aeruginosa | 1 |

29. Secondary Outcome: Composite Success in Patients With Cefepime-Resistant Pathogens at Test of Cure (TOC) in the ME Population
Description: as for outcome 4
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 58 | 24
Participants
  Cefepime-resistant Enterobacterales: number analyzed (Participants) | 57 | 24
  Cefepime-resistant Enterobacterales | 44 | 12
  Cefepime-resistant Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Cefepime-resistant Pseudomonas aeruginosa | 0 |

30. Secondary Outcome: Microbiologic Success in Patients With Cefepime-Resistant Pathogens at Test of Cure (TOC) in the ME Population
Description: as for outcome 2
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 58 | 24
Participants
  Cefepime-resistant Enterobacterales: number analyzed (Participants) | 57 | 24
  Cefepime-resistant Enterobacterales | 46 | 14
  Cefepime-resistant Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Cefepime-resistant Pseudomonas aeruginosa | 0 |

31. Secondary Outcome: Composite Success in Cefepime-Resistant Pathogens at Late Follow Up (LFU) in the ME Population
Description: as for outcome 4
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 60 | 26
Participants
  Cefepime-resistant Enterobacterales: number analyzed (Participants) | 59 | 26
  Cefepime-resistant Enterobacterales | 44 | 11
  Cefepime-resistant Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Cefepime-resistant Pseudomonas aeruginosa | 0 |
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 14.0, 95% CI 2-sided [3.8 to 24.3]

32. Secondary Outcome: Microbiologic Success in Cefepime-Resistant Pathogens at Late Follow Up (LFU) in the ME Population
Description: as for outcome 2
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 60 | 26
Participants
  Cefepime-resistant Enterobacterales: number analyzed (Participants) | 59 | 26
  Cefepime-resistant Enterobacterales | 45 | 14
  Cefepime-resistant Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Cefepime-resistant Pseudomonas aeruginosa | 0 |

33. Secondary Outcome: Clinical Success at End of Treatment (EOT) in the Clinically Evaluable (CE) Population
Description: Symptomatic clinical success is defined as symptomatic resolution or return to pre-morbid baseline of all UTI-core symptoms and patient is alive, and patient has not received additional antibacterial therapy for cUTI.
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: The CE analysis population consists of all patients in the ITT analysis population who had a diagnosis of cUTI; received treatment for ≥48 hours; were evaluated at EOT with a response that was not indeterminate; did not violate prior antibacterials exclusion or received concomitant antibiotic therapy with activity against baseline pathogens except for patients failing study drug; or had other confounding factors that interfered with the assessment of outcome including unblinding.
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 425 | 211
Participants | 384 | 187
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 1.7, 95% CI 2-sided [-3.1 to 7.3]

34. Secondary Outcome: Clinical Success at Test of Cure (TOC) in the CE Population
Description: as for outcome 33
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 392 | 196
Participants | 343 | 162
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 4.8, 95% CI 2-sided [-1.1 to 11.5]

35. Secondary Outcome: Clinical Success at Late Follow Up (LFU) in the CE Population
Description: as for outcome 33
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 387 | 190
Participants | 321 | 142
Statistical Analysis 1: Comparison: Cefepime/VNRX-5133 (Taniborbactam) vs Meropenem; Test type: Other; Miettinen and Nurminen = 8.2, 95% CI 2-sided [1.2 to 15.7]

36. Secondary Outcome: Clinical Success in Patients With Cefepime-Resistant Pathogens at End of Treatment (EOT) in the CE Population
Description: as for outcome 33
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 76 | 35
Participants
  Enterobacterales: number analyzed (Participants) | 70 | 33
  Enterobacterales | 63 | 31
  Pseudomonas aeruginosa: number analyzed (Participants) | 6 | 2
  Pseudomonas aeruginosa | 6 | 2

37. Secondary Outcome: Clinical Success in Patients With Cefepime-Resistant Pathogens at Test of Cure (TOC) in the CE Population
Description: as for outcome 33
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 70 | 30
Participants
  Enterobacterales: number analyzed (Participants) | 64 | 28
  Enterobacterales | 56 | 23
  Pseudomonas aeruginosa: number analyzed (Participants) | 6 | 2
  Pseudomonas aeruginosa | 4 | 2

38. Secondary Outcome: Clinical Success in Patients With Cefepime-Resistant Pathogens at Late Follow Up (LFU) in the CE Population
Description: as for outcome 33
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 70 | 30
Participants
  Enterobacterales: number analyzed (Participants) | 65 | 29
  Enterobacterales | 52 | 19
  Pseudomonas aeruginosa: number analyzed (Participants) | 5 | 1
  Pseudomonas aeruginosa | 3 | 1

39. Secondary Outcome: Per-Pathogen Microbiologic Eradication at End of Treatment (EOT) in the microITT Population
Description: Per-pathogen eradication by baseline gram-negative pathogens. The number analyzed corresponds to the number of specified pathogens. The number is the percent of the specified pathogen identified at baseline in each treatment group that had been eradicated.
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: as for outcome 1
Measure: Count of Units; unit: pathogens
Units Other Than Participants: pathogens
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 293 | 143
Number analyzed (pathogens) | 297 | 147
pathogens
  Citrobacter freundii complex: number analyzed (pathogens) | 2 | 2
  Citrobacter freundii complex | 2 | 2
  Citrobacter koseri: number analyzed (pathogens) | 1 | 1
  Citrobacter koseri | 1 | 1
  Enterobacter cloacae complex: number analyzed (pathogens) | 14 | 3
  Enterobacter cloacae complex | 14 | 3
  Escherichia coli: number analyzed (pathogens) | 202 | 99
  Escherichia coli | 197 | 95
  Klebsiella aerogenes: number analyzed (pathogens) | 1 | 1
  Klebsiella aerogenes | 1 | 1
  Klebsiella oxytoca: number analyzed (pathogens) | 5 | 1
  Klebsiella oxytoca | 5 | 1
  Klebsiella pneumoniae: number analyzed (pathogens) | 40 | 20
  Klebsiella pneumoniae | 37 | 20
  Klebsiella variicola: number analyzed (pathogens) | 1 | 1
  Klebsiella variicola | 1 | 1
  Kluyvera ascorbata: number analyzed (pathogens) | 1 | 0
  Kluyvera ascorbata | 1 |
  Morganella morganii: number analyzed (pathogens) | 2 | 2
  Morganella morganii | 2 | 2
  Proteus hauseri: number analyzed (pathogens) | 1 | 0
  Proteus hauseri | 1 |
  Proteus mirabilis: number analyzed (pathogens) | 10 | 10
  Proteus mirabilis | 10 | 10
  Proteus penneri: number analyzed (pathogens) | 1 | 0
  Proteus penneri | 1 |
  Proteus vulgaris: number analyzed (pathogens) | 2 | 0
  Proteus vulgaris | 2 |
  Serratia marcescens: number analyzed (pathogens) | 2 | 0
  Serratia marcescens | 2 |
  Providencia rettgeri: number analyzed (pathogens) | 0 | 1
  Providencia rettgeri |  | 1
  Pseudomonas aeruginosa: number analyzed (pathogens) | 12 | 6
  Pseudomonas aeruginosa | 11 | 6

40. Secondary Outcome: Per-Pathogen Microbiologic Eradication at Test of Cure (TOC) in the microITT Population
Description: as for outcome 39
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: as for outcome 1
Measure: Count of Units; unit: pathogens
Units Other Than Participants: pathogens
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 293 | 143
Number analyzed (pathogens) | 297 | 147
pathogens
  Citrobacter freundii complex: number analyzed (pathogens) | 2 | 2
  Citrobacter freundii complex | 2 | 2
  Citrobacter koseri: number analyzed (pathogens) | 1 | 1
  Citrobacter koseri | 0 | 1
  Enterobacter cloacae complex: number analyzed (pathogens) | 14 | 3
  Enterobacter cloacae complex | 12 | 1
  Escherichia coli: number analyzed (pathogens) | 202 | 99
  Escherichia coli | 165 | 67
  Klebsiella aerogenes: number analyzed (pathogens) | 1 | 1
  Klebsiella aerogenes | 0 | 0
  Klebsiella oxytoca: number analyzed (pathogens) | 5 | 1
  Klebsiella oxytoca | 5 | 1
  Klebsiella pneumoniae: number analyzed (pathogens) | 40 | 20
  Klebsiella pneumoniae | 27 | 14
  Klebsiella varricola: number analyzed (pathogens) | 1 | 1
  Klebsiella varricola | 1 | 1
  Kluyvera ascorbata: number analyzed (pathogens) | 1 | 0
  Kluyvera ascorbata | 1 |
  Morganella morganii: number analyzed (pathogens) | 2 | 2
  Morganella morganii | 2 | 2
  Proteus hauseri: number analyzed (pathogens) | 1 | 0
  Proteus hauseri | 0 |
  Proteus mirabilis: number analyzed (pathogens) | 10 | 10
  Proteus mirabilis | 9 | 5
  Proteus penneri: number analyzed (pathogens) | 1 | 0
  Proteus penneri | 1 |
  Proteus vulgaris: number analyzed (pathogens) | 2 | 0
  Proteus vulgaris | 1 |
  Providencia rettgeri: number analyzed (pathogens) | 0 | 1
  Providencia rettgeri |  | 1
  Serratia marcescens: number analyzed (pathogens) | 2 | 0
  Serratia marcescens | 2 |
  Pseudomonas aeruginosa: number analyzed (Participants) | 293 | 6
  Pseudomonas aeruginosa: number analyzed (pathogens) | 12 | 6
  Pseudomonas aeruginosa | 5 | 4

41. Secondary Outcome: Per-Pathogen Microbiologic Eradication at Late Follow Up (LFU) in the microITT Population
Description: as for outcome 39
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: as for outcome 1
Measure: Count of Units; unit: pathogens
Units Other Than Participants: pathogens
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 293 | 143
Number analyzed (pathogens) | 297 | 147
pathogens
  Citrobacter freundii complex: number analyzed (pathogens) | 2 | 2
  Citrobacter freundii complex | 1 | 2
  Citrobacter koseri: number analyzed (pathogens) | 1 | 1
  Citrobacter koseri | 0 | 1
  Enterobacter cloacae complex: number analyzed (pathogens) | 14 | 3
  Enterobacter cloacae complex | 12 | 1
  Escherichia coli: number analyzed (pathogens) | 202 | 99
  Escherichia coli | 141 | 61
  Klebsiella aerogenes: number analyzed (pathogens) | 1 | 1
  Klebsiella aerogenes | 0 | 0
  Klebsiella oxytoca: number analyzed (pathogens) | 5 | 1
  Klebsiella oxytoca | 4 | 1
  Klebsiella pneumoniae: number analyzed (pathogens) | 40 | 20
  Klebsiella pneumoniae | 30 | 14
  Klebsiella variicola: number analyzed (pathogens) | 1 | 1
  Klebsiella variicola | 1 | 1
  Kluyvera ascorbata: number analyzed (pathogens) | 1 | 0
  Kluyvera ascorbata | 1 |
  Morganella morganii: number analyzed (pathogens) | 2 | 2
  Morganella morganii | 2 | 2
  Proteus hauseri: number analyzed (pathogens) | 1 | 0
  Proteus hauseri | 0 |
  Proteus mirabilis: number analyzed (pathogens) | 10 | 10
  Proteus mirabilis | 8 | 6
  Proteus penneri: number analyzed (pathogens) | 1 | 0
  Proteus penneri | 1 |
  Proteus vulgaris: number analyzed (pathogens) | 2 | 0
  Proteus vulgaris | 2 |
  Providencia rettgeri: number analyzed (pathogens) | 0 | 1
  Providencia rettgeri |  | 1
  Serratia marcescens: number analyzed (pathogens) | 2 | 0
  Serratia marcescens | 2 |
  Pseudomonas aeruginosa: number analyzed (pathogens) | 12 | 6
  Pseudomonas aeruginosa | 5 | 4

42. Secondary Outcome: Per-Pathogen Microbiologic Eradication in Patients With Cefepime-Resistant Pathogens at End of Treatment (EOT) in the microITT Population
Description: Per-pathogen eradication by baseline gram-negative pathogens (only pathogens identified 10 or more times are reported). The number analyzed corresponds to the number of specified pathogens. The number is the percent of the specified pathogen identified at baseline in each treatment group that had been eradicated.
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of pathogen eradication
Units Other Than Participants: Pathogens
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 67 | 30
Number analyzed (Pathogens) | 67 | 30
percentage of pathogen eradication
  Enterobacter cloacae complex: number analyzed (Participants) | 6 | 2
  Enterobacter cloacae complex: number analyzed (Pathogens) | 6 | 2
  Enterobacter cloacae complex | 100 | 100
  Escherichia coli: number analyzed (Participants) | 37 | 18
  Escherichia coli: number analyzed (Pathogens) | 37 | 18
  Escherichia coli | 100 | 88.9
  Klebsiella oxytoca: number analyzed (Participants) | 1 | 0
  Klebsiella oxytoca: number analyzed (Pathogens) | 1 | 0
  Klebsiella oxytoca | 100 |
  Klebsiella pneumoniae: number analyzed (Participants) | 20 | 7
  Klebsiella pneumoniae: number analyzed (Pathogens) | 20 | 7
  Klebsiella pneumoniae | 95.0 | 100
  Morganella morganii: number analyzed (Participants) | 0 | 1
  Morganella morganii: number analyzed (Pathogens) | 0 | 1
  Morganella morganii |  | 100
  Proteus mirabilis: number analyzed (Participants) | 2 | 2
  Proteus mirabilis: number analyzed (Pathogens) | 2 | 2
  Proteus mirabilis | 100 | 100
  Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Pseudomonas aeruginosa: number analyzed (Pathogens) | 1 | 0
  Pseudomonas aeruginosa | 100 |

43. Secondary Outcome: Per-Pathogen Microbiologic Eradication in Patients With Cefepime-Resistant Pathogens at Test of Cure (TOC) in the microITT Population
Description: as for outcome 42
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: as for outcome 1
Measure: Number; unit: percentage of eradicated pathogens
Units Other Than Participants: pathogens
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 67 | 30
Number analyzed (pathogens) | 67 | 30
percentage of eradicated pathogens
  Enterobacter cloacae complex: number analyzed (Participants) | 6 | 2
  Enterobacter cloacae complex: number analyzed (pathogens) | 6 | 2
  Enterobacter cloacae complex | 100 | 50.0
  Escherichia coli: number analyzed (Participants) | 37 | 18
  Escherichia coli: number analyzed (pathogens) | 37 | 18
  Escherichia coli | 81.1 | 61.1
  Klebsiella oxytoca: number analyzed (Participants) | 1 | 0
  Klebsiella oxytoca: number analyzed (pathogens) | 1 | 0
  Klebsiella oxytoca | 100 |
  Klebsiella pneumoniae: number analyzed (Participants) | 20 | 7
  Klebsiella pneumoniae: number analyzed (pathogens) | 20 | 7
  Klebsiella pneumoniae | 60.0 | 71.4
  Morganella morganii: number analyzed (Participants) | 0 | 1
  Morganella morganii: number analyzed (pathogens) | 0 | 1
  Morganella morganii |  | 100
  Proteus mirabilis: number analyzed (Participants) | 2 | 2
  Proteus mirabilis: number analyzed (pathogens) | 2 | 2
  Proteus mirabilis | 50.0 | 0
  Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Pseudomonas aeruginosa: number analyzed (pathogens) | 1 | 0
  Pseudomonas aeruginosa | 0 |

44. Secondary Outcome: Per-Pathogen Microbiologic Eradication in Patients With Cefepime-Resistant Pathogens at Late Follow Up (LFU) in the microITT Population
Description: as for outcome 42
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: as for outcome 1
Measure: Number; unit: percentage of pathogen eradication
Units Other Than Participants: pathogens
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 67 | 30
Number analyzed (pathogens) | 67 | 30
percentage of pathogen eradication
  Enterobacter cloacae complex: number analyzed (Participants) | 6 | 2
  Enterobacter cloacae complex: number analyzed (pathogens) | 6 | 2
  Enterobacter cloacae complex | 100 | 50.0
  Escherichia coli: number analyzed (Participants) | 37 | 18
  Escherichia coli: number analyzed (pathogens) | 37 | 18
  Escherichia coli | 73.0 | 50.0
  Klebsiella oxytoca: number analyzed (Participants) | 1 | 0
  Klebsiella oxytoca: number analyzed (pathogens) | 1 | 0
  Klebsiella oxytoca | 100 |
  Klebsiella pneumoniae: number analyzed (Participants) | 20 | 7
  Klebsiella pneumoniae: number analyzed (pathogens) | 20 | 7
  Klebsiella pneumoniae | 65.0 | 71.4
  Morganella morganii: number analyzed (Participants) | 0 | 1
  Morganella morganii: number analyzed (pathogens) | 0 | 1
  Morganella morganii |  | 100
  Proteus mirabilis: number analyzed (Participants) | 2 | 2
  Proteus mirabilis: number analyzed (pathogens) | 2 | 2
  Proteus mirabilis | 50.0 | 0
  Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Pseudomonas aeruginosa: number analyzed (pathogens) | 1 | 0
  Pseudomonas aeruginosa | 0 |

45. Secondary Outcome: Per-Pathogen Microbiologic Eradication at End of Treatment (EOT) in the ME Population
Description: as for outcome 39
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: as for outcome 21
Measure: Count of Units; unit: pathogens
Units Other Than Participants: pathogens
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 282 | 137
Number analyzed (pathogens) | 286 | 141
pathogens
  Citrobacter freundii complex: number analyzed (pathogens) | 2 | 2
  Citrobacter freundii complex | 2 | 2
  Citrobacter koseri: number analyzed (pathogens) | 1 | 1
  Citrobacter koseri | 1 | 1
  Enterobacter cloacae complex: number analyzed (pathogens) | 14 | 3
  Enterobacter cloacae complex | 14 | 3
  Escherichia coli: number analyzed (pathogens) | 195 | 94
  Escherichia coli | 193 | 94
  Klebsiella aerogenes: number analyzed (pathogens) | 1 | 1
  Klebsiella aerogenes | 1 | 1
  Klebsiella oxytoca: number analyzed (pathogens) | 5 | 1
  Klebsiella oxytoca | 5 | 1
  Klebsiella pneumoniae: number analyzed (pathogens) | 38 | 20
  Klebsiella pneumoniae | 37 | 20
  Klebsiella variicola: number analyzed (pathogens) | 1 | 1
  Klebsiella variicola | 1 | 1
  Kluyvera ascorbata: number analyzed (pathogens) | 1 | 0
  Kluyvera ascorbata | 1 |
  Morganella morganii: number analyzed (pathogens) | 2 | 2
  Morganella morganii | 2 | 2
  Proteus hauseri: number analyzed (pathogens) | 1 | 0
  Proteus hauseri | 1 |
  Proteus mirabilis: number analyzed (pathogens) | 9 | 9
  Proteus mirabilis | 9 | 9
  Proteus penneri: number analyzed (pathogens) | 1 | 0
  Proteus penneri | 1 |
  Proteus vulgaris: number analyzed (pathogens) | 2 | 0
  Proteus vulgaris | 2 |
  Providencia rettgeri: number analyzed (pathogens) | 0 | 1
  Providencia rettgeri |  | 1
  Serratia marcescens: number analyzed (pathogens) | 2 | 0
  Serratia marcescens | 2 |
  Pseudomonas aeruginosa: number analyzed (pathogens) | 11 | 6
  Pseudomonas aeruginosa | 11 | 6

46. Secondary Outcome: Per-Pathogen Microbiologic Eradication at Test of Cure (TOC) in the ME Population
Description: as for outcome 39
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: as for outcome 23
Measure: Count of Units; unit: pathogens
Units Other Than Participants: pathogens
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 261 | 127
Number analyzed (pathogens) | 265 | 131
pathogens
  Citrobacter freundii complex: number analyzed (pathogens) | 2 | 2
  Citrobacter freundii complex | 2 | 2
  Citrobacter koseri: number analyzed (pathogens) | 0 | 1
  Citrobacter koseri | 0 | 1
  Enterobacter cloacae complex: number analyzed (pathogens) | 13 | 2
  Enterobacter cloacae complex | 11 | 0
  Escherichia coli: number analyzed (pathogens) | 181 | 89
  Escherichia coli | 154 | 64
  Klebsiella aerogenes: number analyzed (pathogens) | 1 | 1
  Klebsiella aerogenes | 0 | 0
  Klebsiella oxytoca: number analyzed (pathogens) | 5 | 1
  Klebsiella oxytoca | 5 | 1
  Klebsiella pneumoniae: number analyzed (pathogens) | 34 | 17
  Klebsiella pneumoniae | 26 | 12
  Klebsiella variicola: number analyzed (pathogens) | 1 | 1
  Klebsiella variicola | 1 | 1
  Kluyvera ascorbata: number analyzed (pathogens) | 1 | 0
  Kluyvera ascorbata | 1 |
  Morganella morganii: number analyzed (pathogens) | 2 | 1
  Morganella morganii | 2 | 1
  Proteus hauseri: number analyzed (pathogens) | 1 | 0
  Proteus hauseri | 0 |
  Proteus mirabilis: number analyzed (pathogens) | 9 | 9
  Proteus mirabilis | 8 | 5
  Proteus penneri: number analyzed (pathogens) | 1 | 0
  Proteus penneri | 1 |
  Proteus vulgaris: number analyzed (pathogens) | 1 | 0
  Proteus vulgaris | 1 |
  Providencia rettgeri: number analyzed (pathogens) | 0 | 1
  Providencia rettgeri |  | 1
  Serratia marcescens: number analyzed (pathogens) | 1 | 0
  Serratia marcescens | 1 |
  Pseudomonas aeruginosa: number analyzed (pathogens) | 12 | 6
  Pseudomonas aeruginosa | 5 | 4

47. Secondary Outcome: Per-Pathogen Microbiologic Eradication at Late Follow Up (LFU) in the ME Population
Description: as for outcome 39
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: as for outcome 25
Measure: Count of Units; unit: pathogens
Units Other Than Participants: pathogens
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 262 | 128
Number analyzed (pathogens) | 266 | 132
pathogens
  Citrobacter freundii complex: number analyzed (pathogens) | 1 | 2
  Citrobacter freundii complex | 1 | 2
  Citrobacter koseri: number analyzed (pathogens) | 0 | 1
  Citrobacter koseri |  | 1
  Enterobacter cloacae complex: number analyzed (pathogens) | 14 | 3
  Enterobacter cloacae complex | 12 | 1
  Escherichia coli: number analyzed (pathogens) | 179 | 86
  Escherichia coli | 130 | 56
  Klebsiella aerogenes: number analyzed (pathogens) | 1 | 1
  Klebsiella aerogenes | 0 | 0
  Klebsiella oxytoca: number analyzed (pathogens) | 4 | 1
  Klebsiella oxytoca | 3 | 1
  Klebsiella pneumoniae: number analyzed (pathogens) | 37 | 19
  Klebsiella pneumoniae | 29 | 14
  Klebsiella variicola: number analyzed (pathogens) | 1 | 1
  Klebsiella variicola | 1 | 1
  Kluyvera ascorbata: number analyzed (pathogens) | 1 | 0
  Kluyvera ascorbata | 1 |
  Morganella morganii: number analyzed (pathogens) | 2 | 1
  Morganella morganii | 2 | 1
  Proteus hauseri: number analyzed (pathogens) | 1 | 0
  Proteus hauseri | 0 |
  Proteus mirabilis: number analyzed (pathogens) | 8 | 10
  Proteus mirabilis | 6 | 6
  Proteus penneri: number analyzed (pathogens) | 1 | 0
  Proteus penneri | 1 |
  Proteus vulgaris: number analyzed (pathogens) | 2 | 0
  Proteus vulgaris | 2 |
  Providencia rettgeri: number analyzed (pathogens) | 0 | 1
  Providencia rettgeri |  | 1
  Serratia marcescens: number analyzed (pathogens) | 2 | 0
  Serratia marcescens | 2 |
  Pseudomonas aeruginosa: number analyzed (pathogens) | 12 | 6
  Pseudomonas aeruginosa | 5 | 4

48. Secondary Outcome: Per-Pathogen Microbiologic Eradication in Patients With Cefepime-Resistant Pathogens at End of Treatment (EOT) in the ME Population
Description: as for outcome 42
Time Frame: Assessed within 24 hours after last IV dose (up to 15 days from start of treatment)
Population: as for outcome 21
Measure: Number; unit: percentage of pathogen eradication
Units Other Than Participants: pathogens
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 64 | 28
Number analyzed (pathogens) | 64 | 28
percentage of pathogen eradication
  Enterobacter cloacae complex: number analyzed (Participants) | 6 | 2
  Enterobacter cloacae complex: number analyzed (pathogens) | 6 | 2
  Enterobacter cloacae complex | 100 | 100
  Escherichia coli: number analyzed (Participants) | 34 | 16
  Escherichia coli: number analyzed (pathogens) | 34 | 16
  Escherichia coli | 100 | 100
  Klebsiella oxytoca: number analyzed (Participants) | 1 | 0
  Klebsiella oxytoca: number analyzed (pathogens) | 1 | 0
  Klebsiella oxytoca | 100 |
  Klebsiella pneumoniae: number analyzed (Participants) | 20 | 7
  Klebsiella pneumoniae: number analyzed (pathogens) | 20 | 7
  Klebsiella pneumoniae | 95.0 | 100
  Morganella morganii: number analyzed (Participants) | 0 | 1
  Morganella morganii: number analyzed (pathogens) | 0 | 1
  Morganella morganii |  | 100
  Proteus mirabilis: number analyzed (Participants) | 2 | 2
  Proteus mirabilis: number analyzed (pathogens) | 2 | 2
  Proteus mirabilis | 100 | 100
  Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Pseudomonas aeruginosa: number analyzed (pathogens) | 1 | 0
  Pseudomonas aeruginosa | 100 |

49. Secondary Outcome: Per-Pathogen Microbiologic Eradication in Patients With Cefepime-Resistant Pathogens at Test of Cure TOC in the ME Population
Description: as for outcome 42
Time Frame: Assessed at Test of Cure visit (occurred once per participant between Study Days 19 to 23)
Population: as for outcome 23
Measure: Number; unit: percentage of pathogen eradication
Units Other Than Participants: Pathogens
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 58 | 24
Number analyzed (Pathogens) | 58 | 24
percentage of pathogen eradication
  Enterobacter cloacae complex: number analyzed (Participants) | 5 | 1
  Enterobacter cloacae complex: number analyzed (Pathogens) | 5 | 1
  Enterobacter cloacae complex | 100 | 0
  Escherichia coli: number analyzed (Participants) | 32 | 15
  Escherichia coli: number analyzed (Pathogens) | 32 | 15
  Escherichia coli | 87.5 | 66.7
  Klebsiella oxytoca: number analyzed (Participants) | 1 | 0
  Klebsiella oxytoca: number analyzed (Pathogens) | 1 | 0
  Klebsiella oxytoca | 100 |
  Klebsiella pneumoniae: number analyzed (Participants) | 17 | 6
  Klebsiella pneumoniae: number analyzed (Pathogens) | 17 | 6
  Klebsiella pneumoniae | 64.7 | 66.7
  Proteus mirabilis: number analyzed (Participants) | 2 | 2
  Proteus mirabilis: number analyzed (Pathogens) | 2 | 2
  Proteus mirabilis | 50.0 | 0
  Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Pseudomonas aeruginosa: number analyzed (Pathogens) | 1 | 0
  Pseudomonas aeruginosa | 0 |

50. Secondary Outcome: Per-Pathogen Microbiologic Eradication in Patients With Cefepime-Resistant Pathogens at Late Follow Up (LFU) in the ME Population
Description: as for outcome 42
Time Frame: Assessed at Late Follow Up visit (occurred once per participant between Study Days 28 to 35)
Population: as for outcome 25
Measure: Number; unit: percentage of pathogen eradication
Units Other Than Participants: pathogens
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 60 | 26
Number analyzed (pathogens) | 60 | 26
percentage of pathogen eradication
  Enterobacter cloacae complex: number analyzed (Participants) | 6 | 2
  Enterobacter cloacae complex: number analyzed (pathogens) | 6 | 2
  Enterobacter cloacae complex | 100 | 50.0
  Escherichia coli: number analyzed (Participants) | 32 | 15
  Escherichia coli: number analyzed (pathogens) | 32 | 15
  Escherichia coli | 78.1 | 53.3
  Klebsiella pneumoniae: number analyzed (Participants) | 19 | 7
  Klebsiella pneumoniae: number analyzed (pathogens) | 19 | 7
  Klebsiella pneumoniae | 68.4 | 71.4
  Proteus mirabilis: number analyzed (Participants) | 2 | 2
  Proteus mirabilis: number analyzed (pathogens) | 2 | 2
  Proteus mirabilis | 50.0 | 0
  Pseudomonas aeruginosa: number analyzed (Participants) | 1 | 0
  Pseudomonas aeruginosa: number analyzed (pathogens) | 1 | 0
  Pseudomonas aeruginosa | 0 |

51. Other Pre Specified Outcome: Number of Patients With Treatment-Emergent Adverse Events
Description: Percent of participants experiencing Treatment Emergent Adverse Events (TEAE). Treatment emergent is defined as any event that starts or worsens during or after treatment.
Time Frame: Study Days 1 to 35
Population: Patients with at least one TEAE.
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 440 | 217
Participants | 156 | 63

52. Other Pre Specified Outcome: Number of Patients With Serious Adverse Events
Description: Percent of participants experiencing treatment emergent Serious Adverse Events (SAE).
Time Frame: Study Days 1 to 35
Population: Patients with at least one treatment-emergent SAE.
Measure: Count of Participants; unit: Participants
Groups:
- Meropenem: Meropenem administered q8h IV over 30 minutes.
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
Number analyzed (Participants) | 440 | 217
Participants | 9 | 4

ADVERSE EVENTS:
Time Frame: From first dose to last follow-up visit (Day 28-35).
Description: Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) in patients who received at least one dose of study drug (Safety Population).
Groups:
- Cefepime/VNRX-5133 (Taniborbactam): Cefepime/VNRX-5133 administered q8h intravenously (IV) over a 2-hour period for 7 days (up to 14 days for patients with bacteremia). Patients also received meropenem placebo administered via IV over a 2-hour period.
- Meropenem: Meropenem administered q8h IV over 30 minutes for 7 days (up to 14 days for patients with bacteremia). Patients also received cefepime/VNRX-5133 placebo administered via IV over a 2-hour period.
Arm/Group | Cefepime/VNRX-5133 (Taniborbactam) | Meropenem
All-Cause Mortality (participants affected / at risk) | 1/440 | 0/217
Serious Adverse Events (participants affected / at risk) | 9/440 | 4/217
Other Adverse Events (participants affected / at risk) | 93/440 | 37/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cefepime/VNRX-5133 (Taniborbactam) (N=440) | Meropenem (N=217)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cefepime/VNRX-5133 (Taniborbactam) (N=440) | Meropenem (N=217)
Headache (Nervous system disorders) | 27 (27) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 18 (18) | 5 (5)
Constipation (Gastrointestinal disorders) | 14 (14) | 3 (3)
Hypertension (Vascular disorders) | 9 (10) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (9) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 7 (7) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 3 (3)
Dizziness (Nervous system disorders) | 7 (7) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 1 (1)
Phlebitis (Vascular disorders) | 6 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Pyrexia (General disorders) | 5 (5) | 3 (3)
Alanine aminotransferase increased (Investigations) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Certain PIs are not allowed to present or publish data from the Study without Sponsor's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT03840148/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT03840148/SAP_001.pdf